CLINICAL TRIAL: NCT01267916
Title: Intrinsic PEEP During Mechanical Ventilation of Patients With Obesity. Influence of Low Respiratory Rate With Unchanged Minute Volume.
Brief Title: Intrinsic PEEP During Mechanical Ventilation of Patients With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul Medical Center (Other)
Responsible Party: Principal Investigator, Won Ho Kim, Staff Anesthesiologist, Seoul Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: SMC-2010-12-13
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: General Anesthesia; Laparoscopic Cholecystectomy
Keywords: intrinsic positive end-expiratory pressure; obesity; ventilator setting; respiratory rate
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (6):
- RR 6 + 0 (Experimental): Respiratory rate 6 Tidal volume 16.7 ml/kg external PEEP = 0
  Interventions: Device: RR 6 + 0
- RR 10 + 0 (Experimental): Respiratory rate 10 Tidal volume 10 ml/kg external PEEP = 0
  Interventions: Device: RR 10 + 0
- RR 16 + 0 (Experimental): Respiratory rate 16 Tidal volume 6.25 ml/kg external PEEP = 0
  Interventions: Device: RR 16 + 0
- RR 6 + 5 (Experimental): Respiratory rate 6 Tidal volume 16.7 ml/kg external PEEP = 5
  Interventions: Device: RR 6 + 5
- RR 10 + 5 (Experimental): Respiratory rate 10 Tidal volume 10 ml/kg external PEEP = 5
  Interventions: Device: RR 10 + 5
- RR 16 + 5 (Experimental): Respiratory rate 16 Tidal volume 6.25 ml/kg external PEEP = 5
  Interventions: Device: RR 16 + 5

INTERVENTIONS:
Device: RR 6 + 0 — Respiratory rate 6 Tidal volume 16.7 ml/kg external PEEP = 0
  Other Names: Ventilator setting
  Arms: RR 6 + 0
Device: RR 10 + 0 — Respiratory rate 10 Tidal volume 10 ml/kg external PEEP = 0
  Other Names: Ventilator setting
  Arms: RR 10 + 0
Device: RR 16 + 0 — Respiratory rate 16 Tidal volume 6.25 ml/kg external PEEP = 0
  Other Names: Ventilator setting
  Arms: RR 16 + 0
Device: RR 6 + 5 — Respiratory rate 6 Tidal volume 16.7 ml/kg external PEEP = 5
  Other Names: Ventilator setting
  Arms: RR 6 + 5
Device: RR 10 + 5 — Respiratory rate 10 Tidal volume 10 ml/kg external PEEP = 5
  Other Names: Ventilator setting
  Arms: RR 10 + 5
Device: RR 16 + 5 — Respiratory rate 16 Tidal volume 6.25 ml/kg external PEEP = 5
  Other Names: Ventilator setting
  Arms: RR 16 + 5

SUMMARY:
It is demonstrated that expiratory flow limitation and as a consequence, intrinsic positive end-expiratory pressure (PEEP) is present in grossly obese subjects especially in the supine position. The investigators tried to investigate the effect of low respiratory rate and high tidal volume on the intrinsic PEEP and gas exchange for obese subjects undergoing general anesthesia.

DETAILED DESCRIPTION:
Impaired gas exchange is a common anesthetic problem in obese subjects. It is demonstrated that expiratory flow limitation and as a consequence, intrinsic positive end-expiratory pressure (PEEPi) is present in grossly obese subjects especially in the supine position. It is known that there is a significant negative correlation between PEEPi present and PaO2. Therefore, the investigators postulated that if the reduce the PEEPi by reducing the respiratory rate in obese subjects, the impaired gas exchange might improve.

The investigators tried to research the effect of low respiratory rate and high tidal volume on the intrinsic PEEP and gas exchange for obese subjects undergoing general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I or II obesity, Body-mass index > 27.5 undergoing laparoscopic cholecystectomy

Exclusion Criteria:

* patients with severe cardiopulmonary disease peak inspiratory pressure > 40 in the study setting

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Gas change parameters | 15 minute interval
  PaO2 and PaCO2 the result of arterial blood gas analysis

SECONDARY OUTCOMES:
intrinsic positive end-expiratory pressure | every 15 minutes
  PEEPi measured by expiratory port occlusion method

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul Medical Center, Seoul, South Korea